CLINICAL TRIAL: NCT05986864
Title: Phase I/II Study to Evaluate the Safety and Preliminary Efficacy of SKG0106 Intravitreal Injection in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Phase I/II Study of SKG0106 Intravitreal Injection in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Skyline Therapeutics (US) Inc. (Industry)
Responsible Party: Sponsor
Organization: Skyline Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKG0106-101
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD; wet AMD; wAMD; nAMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I: Low dose (Experimental): SKG0106 One-Time Intraocular Injection Dose Level 1
  Interventions: Genetic: SKG0106
- Phase I: Medium dose (Experimental): SKG0106 One-Time Intraocular Injection Dose Level 2
  Interventions: Genetic: SKG0106
- Phase I: High dose (Experimental): SKG0106 One-Time Intraocular Injection Dose Level 3
  Interventions: Genetic: SKG0106

INTERVENTIONS:
Genetic: SKG0106 — SKG0106 is a recombinant adeno-associated virus (AAV) vector-based in vivo gene therapeutic product

SUMMARY:
This is a phase 1/2 clinical study to evaluate the safety, preliminary efficacy, immunogenicity, and pharmacokinetic (PK) characteristics of SKG0106 in subjects with nAMD. Based on results from the phase 1 dose escalation study, the phase 2 expansion study will be conducted.

ELIGIBILITY:
Inclusion criteria:

1. Voluntary and able to sign a dated ICF prior to any study-related procedures and able to complete the study as required by the protocol;
2. Aged ≥ 50 years at screening;

   Study Eye:
3. Diagnosis of nAMD as determined by the PI;
4. Active CNV lesions secondary to age-related macular degeneration (AMD);
5. Subjects must have been responsive to anti-VEGF therapy as assessed by the PI prior to study treatment.

Exclusion Criteria:

1. Any active intraocular or periocular infection or active intraocular inflammation (e.g., infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in the study eye at baseline;
2. Retinal pigment epithelial tear in the study eye at screening;
3. Current vitreous hemorrhage in the study eye or history of vitreous hemorrhage within 4 weeks prior to baseline;
4. Any condition that, in the opinion of the investigator, may limit visual acuity improvement in the study eye;
5. History of retinal detachment or active retinal detachment in the study eye;
6. Any prior gene therapy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Characteristics of dose limiting toxicities (DLTs) | 4 Weeks
Type, severity, and incidence of ocular and systemic adverse events (AEs) | 52 Weeks

SECONDARY OUTCOMES:
Mean change from baseline in best corrected visual acuity (BCVA) at each visit | 52 Weeks
  BCVA of the study eye is examined by the Early Treatment of Diabetic Retinopathy Study (ETDRS) testing at screening and baseline.
Mean change from baseline in central subfield thickness (CST) at each visit | 52 Weeks
  Spectral domain optical coherence tomography (SD-OCT) will be performed to measure CST at screening and at each visit (prior to study drug injection, if available).
Mean change from baseline in patient-reported outcome (VFQ-25) scale score at each visit | 52 Weeks
  Both the total scale and subscale scores of the VFQ-25 is ranging from 0 to 100, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Retina Vitreous Associates of Florida - Saint Petersburg, St. Petersburg, Florida
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Texas, Katy, Texas
  - Wagner Kapoor Research Institute, Norfolk, Virginia
- China (5):
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Eye Hospital, WMU (Zhejiang Eye Hospital), Wenzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No